CLINICAL TRIAL: NCT01713114
Title: A Randomized, Controlled Crossover Trial to Assess the Effects of Varying Meals on Satiety
Brief Title: Effects of a Variety of Meals on Satiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hillshire Brands Company (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: PRV1223
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Focus of the Study is Satiety

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (4):
- Low carbohydrate (Experimental)
  Interventions: Other: Acute measures of satiety and food intake at next meal
- Moderate carbohydrate (Experimental)
  Interventions: Other: Acute measures of satiety and food intake at next meal
- Higher Carbohydrate (Experimental)
  Interventions: Other: Acute measures of satiety and food intake at next meal
- Meal Skipping (Placebo Comparator)
  Interventions: Other: Acute measures of satiety and food intake at next meal

INTERVENTIONS:
Other: Acute measures of satiety and food intake at next meal

SUMMARY:
The primary objective of this study is to assess the acute effects of different meals on satiety. It is hypothesized that a lower carbohydrate meal will result in greater feelings of satiety and reduced food intake at a subsequent meal compared to the higher-carbohydrate or meal skipping conditions.

DETAILED DESCRIPTION:
Satiety refers to feelings of fullness or lack of desire to eat following consumption of a food or meal. A number of dietary factors have been shown to influence satiety, including food volume, food weight, energy density, food palatability, and certain food ingredients. The nutritional composition of a meal appears to also play a significant role in an individual's feelings of satiety and ability to stay full until the next meal.

ELIGIBILITY:
Inclusion Criteria:

* premenopausal Females
* Ages 18-55
* BMI between 18.5-29.9
* Willing to maintain weight throughout study period

Exclusion Criteria:

* Subject has a history of any surgical intervention for the treatment of obesity
* Recent history or use of weight loss drugs, herbal supplements or on a dieting program or trying to loose weight
* Gains or loses more than 6 pounds over the study period
* Current or history of an eating disorder
* Restrained eater
* Excludes any foods or meals from their diet
* History or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, gastrointestinal, biliary, pancreatic or neurologic disorders
* Signs of an infection
* Heavy user of caffeine or alcohol
* Unconventional sleep patterns (e.g. works 3rd shift)
* Subject is pregnant or planning to become pregnant during the study period

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Composite Area under the Curve - Visual Analog Scale | Acute - up to 4 hrs

SECONDARY OUTCOMES:
Individual satiety measures - Area under the curve | 4 hrs

OTHER OUTCOMES:
Differences between test conditions in food intake, energy intake and areas under the curve. | 4 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis Clinical Research, Addison, Illinois, United States

REFERENCES:
- [Derived] Rains TM, Leidy HJ, Sanoshy KD, Lawless AL, Maki KC. A randomized, controlled, crossover trial to assess the acute appetitive and metabolic effects of sausage and egg-based convenience breakfast meals in overweight premenopausal women. Nutr J. 2015 Feb 10;14:17. doi: 10.1186/s12937-015-0002-7. PMID 25889354